CLINICAL TRIAL: NCT01000714
Title: Determination of the Efficacy and Safety of Psirelax in the Relief of the Disease in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Etwal Ltd. (Industry)
Other Study IDs: protocol No. 1 ver. 1 9-Jan-09
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Mild to Moderate Psoriasis

INTERVENTIONS:
Drug: Psirelax

SUMMARY:
Psoriasis is a chronic disorder characterized by erythematous scaly patches which affect the scalp, trunk, extensor surfaces of the limbs and the genital area. The common form of psoriasis is referred to as psoriasis vulgaris. There are several variants of psoriasis such as guttate psoriasis, inverse psoriasis, pustular psoriasis and erythrodermic psoriasis.

Psoriasis is highly prevalent in the general population, mainly as a result of its chronicity and the absence of a cure. The estimates of psoriasis prevalence are within the range of 0.5% to 4%.

The diagnosis of psoriasis is made on a clinical base, usually by physical examination, performed by a dermatologist. Although skin biopsy may be useful in some cases, there is no laboratory test which may serve as a reference standard to the clinical diagnosis of psoriasis.

Psoriasis in its mild cases per se is not associated with excess mortality, however, the disease may affect quality of life of affected patients to a substantial degree. Psoriasis may be readily apparent to others because of scales and redness of the skin. The skin may itch and scales may shed from the patients to the environment or directly on other people. Feelings of stigmatization and major changes in life-style caused by psoriasis have been documented in numerous studies. The burden of the disease may be exaggerated due to expensive therapy and complicated therapeutic regimes Patients with mild to moderate psoriasis are usually treated with topical treatments. Photo-therapy or systemic treatments are reserved to patients with moderate to severe disease.

Topical corticosteroids may lead to rapid improvement in psoriasis, however rapid relapse following discontinuation is the common practice leading to chronic use.

Calcipotriene ointment may also be used and requires 8 to 12 weeks of use for maximal effect and often causes local irritation, particularly when used on the face. The use is limited to 100 gr/week due to hypercalcemia that might follow systemic absorption.

Vitamin A derivative tazarotene may be also be used for plaque psoriasis. Although it can produce longer remissions than topical steroids, local irritation, cost, and teratogenicity limit its use.

Coal tar products may be used as steroid-sparing agents, especially useful for enhancing the efficacy of natural sunlight and phototherapy. Application can be cumbersome because of irritation, unpleasant smell, brown color that can stain clothing, and propensity to cause folliculitis.

All of the above treatments are particularly problematic for the face and genital psoriasis due to the potential side effects and mainly possible severe irritation reducing patients compliance.

Psirelax is a novel topical medication directed for the treatment of patients with psoriasis. The formulation of Psirelax includes the following substances: 5%-15% quince seeds jelly, 10%-40% natural base cream (e.g. Ferntree Cottage Pure Base Cream), 55%-75% mixture of natural anti-oxidants (e.g. Vitamin E, wheat germ oil, Safflower oil), natural skin softening agents (e.g. sweet almond oil, sesame oil), natural absorption aids (e.g. jojoba oil, vegetable squalene), natural tissue regenerating and protecting agents (e.g. grape seed oil, sunflower oil), natural preservatives (e.g. paraben, tea trea essential oil, thyme essential oil, grapefruit seed extract, Vitamin E) and natural thickening agents (e.g. bee wax, aloevera, medicinal Vaseline, coconut oil, guar gum, palm oil, borax)

In a preliminary observation, a patient with severe psoriasis applied Psirelax three times each day during four days. The patient reported complete disappearance of the psoriatic plaques and pruritus was reduced by 70%. It was suggested to conduct an open study to assess the effect of Psirelax in patients with psoriasis vulgaris.

The aim of this study is to examine the safety and efficacy of Psirelax in the treatment of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 18 and 75 years old, inclusive.
2. Clinical diagnosis of psoriasis.
3. In otherwise good general health and free of any disease or physical condition which might impair evaluation of plaque psoriasis.
4. Able to understand and willing to comply with all study requirements, particularly the regimen for administration of study drug.
5. Able to understand and willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Women who are pregnant, lactating, planning to become pregnant, or women of child-bearing potential who have not successfully been using the same medically acceptable contraceptive methods over the previous 3 months, e.g., oral contraceptive agents, intrauterine device (IUD), and barrier method plus spermicide.
2. Use of topical anti psoriatic therapy (including topical retinoids, corticosteroids, or vitamin D analogs) on the areas to be treated within one week prior to the beginning of the study.
3. Received systemic biologic therapy to treat psoriasis (e.g., alefacept, etanercept, infliximab, efalizumab, adalimumab) within 12 weeks prior to the beginning of the study.
4. Received systemic psoriasis therapy (e.g., methotrexate, cyclosporine, systemic corticosteroids, retinoids such as acitretin) within 4 weeks prior to the beginning of the study.
5. Received phototherapy (including laser), photo chemotherapy for the study areas within 4 weeks prior to the beginning of the study.
6. Recent history (within past 12 months) of alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 4 oz wine, or 1.5 oz distilled spirits).
7. History of noncompliance to medical regimens or unwilling to comply with the study protocol.
8. Participation in an investigational drug study within 30 days prior to the beginning of the study.
9. Serious or unstable medical or psychological conditions that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Clalit Health care, Tel Aviv, Israel